CLINICAL TRIAL: NCT07378709
Title: Blood-Based Biomarkers for Prediction and Monitoring of Response to TACE in Hepatocellular Carcinoma: A Pilot Study
Brief Title: Exploratory Blood-Based Biomarkers in TACE-Treated Hepatocellular Carcinoma
Acronym: BLOOD-TACE-P
Status: Recruiting | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Marko Stojanovic, Associate Professor, Department of Pharmacology, Clinical Pharmacology and Toxicology, University of Belgrade
Other Study IDs: 6249_pilot_study
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma (HCC); Liver Neoplasms
Keywords: Hepatocellular Carcinoma; TACE; Biomarkers; mRECIST; Drug-Eluting Beads
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (serum and plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC Patients Treated With TACE: Patients with hepatocellular carcinoma (HCC) who are candidates for transarterial chemoembolization (TACE) as part of their standard clinical care. This group includes adult patients with preserved liver function (Child-Pugh ≤ 7) and good performance status Eastern Cooperative Oncology Group (ECOG) 0.

SUMMARY:
The goal of this observational study is to evaluate changes in selected biomarkers and their potential connection with early radiological outcomes in adult patients with hepatocellular carcinoma (HCC) who are candidates for Transarterial Chemoembolization (TACE) treatment. The main questions it aims to answer are whether specific biomarkers change in response to TACE treatment and if there is a correlation between these changes and early radiological treatment response as measured by Modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria. Participants will undergo standard-of-care TACE as decided by a multidisciplinary team and will provide blood samples at predefined, clinically relevant time points, specifically before the first TACE procedure and during subsequent follow-up cycles on the day of either a new TACE or a control Computed Tomography (CT) scan. Additionally, participants will undergo routine clinical and radiological assessments, including multiphase CT or Magnetic Resonance Imaging (MRI) scans four to eight weeks after the procedure to monitor treatment success, with all data being collected from medical records and standard diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of hepatocellular carcinoma (HCC) based on LI-RADS CT/MRI v2018 criteria or histopathological verification
* Candidate for TACE as part of standard treatment (BCLC criteria)
* Child-Pugh score ≤ 7 at the time of TACE indication
* ECOG performance status 0 at the time of TACE indication
* Availability of at least one follow-up multiphase CT or MRI scan 4-8 weeks after TACE

Exclusion Criteria:

* Child-Pugh score ≥8 at the time of TACE indication
* Eastern Cooperative Oncology Group (ECOG) performance status > 0 at the time of TACE indication.
* Presence of extrahepatic dissemination and/or macrovascular invasion
* Technically unfeasible TACE (e.g., inability to identify feeder artery)
* Severe uncorrectable coagulopathy or cytopenia
* Severe allergy or contraindication to iodine contrast agent or drugs used during TACE
* Pregnancy or breastfeeding
* Inability to provide signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma (HCC) treated with transarterial chemoembolization (TACE) at the University Hospital Center (KBC) Bežanijska kosa
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between blood-based biomarkers and early radiological response | From baseline (before first TACE) up to the follow-up assessment 4-8 weeks after the procedure.
  Evaluation of changes in selected biomarkers (including AFP and PIVKA-II) and their potential association with early radiological outcomes following TACE, assessed using mRECIST criteria (Complete Response, Partial Response, Stable Disease, or Progressive Disease).

SECONDARY OUTCOMES:
Radiological Response Assessment via mRECIST. | 4-8 weeks after each TACE procedure.
  Tumor response will be evaluated according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST), a categorical scale used to assess viable tumor based on arterial enhancement on CT or MRI scans.
  Scale Information:
  Scale Type: Categorical
  Minimum Value: Complete Response (CR) - best outcome
  Maximum Value: Progressive Disease (PD) - worst outcome
  Directionality: Higher category represents a worse outcome
  Categories:
  Complete Response (CR)
  Partial Response (PR)
  Stable Disease (SD)
  Progressive Disease (PD)
  Outcome Reporting:
  The percentage of patients achieving each response category (CR, PR, SD, PD) will be reported.
Changes in Tumor Marker Levels (AFP and PIVKA-II). | Baseline (Day 0, before first TACE) and at each follow-up cycle (4-8 weeks after procedure).
  Measurement of the change in serum levels of Alpha-fetoprotein (AFP) and Protein Induced by Vitamin K Absence (PIVKA-II from baseline to follow-up points.
Assessment of Liver Function Post-TACE. | From baseline up to 8 weeks after the final TACE procedure.
  Liver function will be monitored using the Child-Pugh Liver Function Score, which evaluates hepatic reserve based on five clinical and laboratory parameters (bilirubin, albumin, INR/prothrombin time, ascites, and hepatic encephalopathy).
  The score is calculated at baseline and during follow-up assessments to evaluate potential liver function deterioration after TACE.
  Scale Information:
  Full Scale Name: Child-Pugh Liver Function Score
  Scale Type: Ordinal numeric scale with clinical class categories
  Minimum Value: 5 points - best liver function (Child-Pugh Class A)
  Maximum Value: 15 points - worst liver function (Child-Pugh Class C)
  Directionality: Higher scores represent a worse clinical outcome
  Score Ranges / Classes:
  5-6 points: Child-Pugh A (well-compensated liver disease)
  7-9 points: Child-Pugh B (significant functional impairment)
  10-15 points: Child-Pugh C (severe hepatic dysfunction)
Exploratory Serum Biomarker Profiling (Proteomics, miRNA, and Oxidative Stress). | From baseline (Day 0, before first TACE) up to the first follow-up assessment (4-8 weeks post-procedure).
  An exploratory evaluation of serum samples to identify changes in protein profiles (proteomics), circulating microRNA (miRNA) signatures, and markers of oxidative stress (e.g., Malondialdehyde, Superoxide Dismutase) as potential predictors or indicators of radiological response to Drug-eluting Bead Trans arterial Chemoembolization (DEB-TACE).

CONTACTS AND LOCATIONS:
Locations (1):
- KBC Bežanijska kosa, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect patient privacy and confidentiality, as the informed consent form signed by participants does not include a provision for the public sharing of raw individual data. Furthermore, as a pilot study, the primary focus is on generating preliminary evidence and internal hypothesis testing.